CLINICAL TRIAL: NCT02345564
Title: Clinical and Radiological Results of Osteochondral Repair Using MaioRegen in Knee and Ankle Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barmherzige Brüder Eisenstadt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBEMaRe 001
Record Dates: First submitted 2014-09-11; First posted 2015-01-26 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Osteochondral Lesion of Talus; Degenerative Lesion of Articular Cartilage of Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- osteochondral lesions in knee/ankle (Other): patients with traumatic and atraumatic osteochondral lesions in knee/ankle, implantation of MaioRegen fleece into osteochondral lesion
  Interventions: Device: implantation of MaioRegen fleece into osteochondral lesion

INTERVENTIONS:
Device: implantation of MaioRegen fleece into osteochondral lesion — arthroscopic localization of lesion, arthroscopic guided mini-arthrotomy and implantation of defect sized MaioRegen fleece
  Other Names: MaioRegen Fin-Ceramica Faenza S.p.A.

SUMMARY:
Osteochondral lesions in knee and ankle are injuries commonly seen in young patients. MaioRegen fleece is a cartilage substitute which can be used in circumscribed defects.

This prospective study follows patients treated with MaioRegen implants from pre-surgery until 24 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* single osteochondral lesion in knee/ankle (2-4 sq cm)

Exclusion Criteria:

* multiple osteochondral lesions
* pre-existing injuries/arthropathies

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
MRI imaging - gap between cartilage-implant surface in mm | 18 months post surgery
  ingrowth of fleece into the cartilage

SECONDARY OUTCOMES:
clinical outcome measurement | pre-surgery
  Lysholm Knee Score Cincinatti Knee Scale IKDC Knee Score AOFAS Hindfoot Score Foot&Ankle Disability Index
clinical outcome measurement | 6 months post-surgery
  Lysholm Knee Score Cincinatti Knee Scale IKDC Knee Score AOFAS Hindfoot Score Foot&Ankle Disability Index
clinical outcome measurement | 12 months post-surgery
  Lysholm Knee Score Cincinatti Knee Scale IKDC Knee Score AOFAS Hindfoot Score Foot&Ankle Disability Index
clinical outcome measurement | 18 months post-surgery
  Lysholm Knee Score Cincinatti Knee Scale IKDC Knee Score AOFAS Hindfoot Score Foot&Ankle Disability Index
clinical outcome measurement | 24 months post-surgery
  Lysholm Knee Score Cincinatti Knee Scale IKDC Knee Score AOFAS Hindfoot Score Foot&Ankle Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kellner, MD, Principal Investigator — Barmherzige Brueder Eisenstadt; Harald Boszotta, MD, Study Chair — Barmherzige Brueder Eisenstadt